CLINICAL TRIAL: NCT00135291
Title: Effect of Leukoreduction in Infection Risk in Trauma
Brief Title: Effect of Leukoreduced Blood Transfusions on Infection Following Trauma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Avery B Nathens, MD PhD MPH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02-2517-D02; P50HL073996-01 (NIH)
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2008-01-11 (Estimated); Status verified 2008-01

CONDITIONS: Wounds and Injuries
Keywords: transfusion-induced immunomodulation; leukoreduction; surgical site infections; nosocomial infections; transfusion; Infection; Sepsis; Hemorrhage
MeSH Terms: conditions — Wounds and Injuries; Surgical Wound Infection; Cross Infection; Infections; Sepsis; Hemorrhage

INTERVENTIONS:
Procedure: Leukoreduced blood transfusion

SUMMARY:
The purpose of this study is to determine if leukoreduced blood transfusions reduce the risk of infection following trauma. Specifically, the investigators intend to evaluate whether there are clinically relevant differences in the rates of infection and in the severity of multiple organ failure in critically injured trauma patients receiving leukoreduced blood products compared to those receiving standard allogeneic blood products.

DETAILED DESCRIPTION:
Many severely injured patients survive their initial resuscitation only to suffer the late sequelae of nosocomial infection and multiple organ failure. The depth of hemorrhagic shock and the severity of anatomic injury are clearly associated with these adverse outcomes, however there is clear evidence to suggest that events during the resuscitation phase also play an important role in the pathogenesis of these sequelae. Specifically, there is now substantial clinical and experimental evidence implicating blood transfusion and the transfusion of allogeneic passenger leukocytes in the immune dysregulation characteristic of the post-injury state. This immune dysregulation manifests on two fronts: an uncontrolled inflammatory response leading to organ dysfunction and a state of immunoparalysis, leading to the development of nosocomial infection. Allogeneic passenger leukocytes have been implicated in the alterations in non-specific and specific immunity that underlie this state of altered immunoresponsiveness. The importance of allogeneic leukocytes in these phenomena suggests that strategies designed to limit the exposure of patients to these cells may reduce the incidence of post-injury sequelae. Pre-storage leukoreduction, whereby donated blood is passed through a leukocyte filter prior to storage and ultimate transfusion is one such strategy. This strategy remains at the center of a national debate on a policy of universal leukoreduction in which its efficacy is unproven and its cost undisputed.

Study Objectives:

* To evaluate whether there are clinically relevant differences in the rates of infection and in the severity of multiple organ failure in critically injured trauma patients receiving leukoreduced blood products compared to those receiving standard allogeneic blood products.
* To assess T-cell responsiveness and the dominant CD4 lymphocyte subset as measured by T-lymphocyte IL-2 receptor expression and cytokine profile, respectively, in critically injured subjects transfused with leukoreduced blood products compared to subjects receiving standard allogeneic blood products.
* To assess the activational state of the peripheral blood monocyte and the neutrophil in critically injured trauma patients receiving leukoreduced blood products compared to subjects receiving standard allogeneic blood products.
* To evaluate whether there are clinically relevant differences in rates of acute lung injury (ALI) and circulating markers of ALI in patients receiving leukoreduced versus standard allogeneic blood products.
* To evaluate rates of microchimerism in those receiving leukoreduced versus standard allogeneic transfusion

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients
* Age > 17
* Transfusion within 24 hours of injury

Exclusion Criteria:

* Active infection at time of injury
* Anticipated survival of < 48 hours (e.g. gunshot wound [GSW] to head, cardiopulmonary resuscitation [CPR] in progress)
* Receipt of blood products for this injury event prior to randomization
* AB negative; B negative blood type.
* Positive antibody screen
* Prior requirement for irradiated, leukoreduced or cytomegalovirus (CMV) seronegative blood products
* Incarcerated
* Enrolled in pre-hospital trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-02; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Infection within 30 days of injury | 30 d

SECONDARY OUTCOMES:
Marshall organ dysfunction scores over the course of Intensive Care Unit (ICU) admission
Hospital length of stay
Duration of mechanical ventilation
Duration of ICU stay
Acute lung injury
Plasma circulating levels of inflammatory cytokines and markers of lung injury (days 2-3 and 6-8)
Measures of monocyte activation (days 2-3 and 6-8)
Measures of polymorphonuclear neutrophil (PMN) activation (days 2-3 and 6-8)
Peripheral blood mononuclear cell expression of interleukin-2 (IL-2) receptors (days 2-3 and 6-8)

CONTACTS AND LOCATIONS:
Overall Officials: Avery B Nathens, MD PhD MPH, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Result] Nathens AB, Nester TA, Rubenfeld GD, Nirula R, Gernsheimer TB. The effects of leukoreduced blood transfusion on infection risk following injury: a randomized controlled trial. Shock. 2006 Oct;26(4):342-7. doi: 10.1097/01.shk.0000228171.32587.a1. PMID 16980879
- [Result] Utter GH, Nathens AB, Lee TH, Reed WF, Owings JT, Nester TA, Busch MP. Leukoreduction of blood transfusions does not diminish transfusion-associated microchimerism in trauma patients. Transfusion. 2006 Nov;46(11):1863-9. doi: 10.1111/j.1537-2995.2006.00991.x. PMID 17076839